CLINICAL TRIAL: NCT04861194
Title: EREctile Function Preservation for Prostate Cancer Radiation Therapy (ERECT); a Prospective Phase II Trial
Brief Title: EREctile Function Preservation for Prostate Cancer Radiation Therapy (ERECT)
Acronym: ERECT
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: UMC Utrecht (Other)
Responsible Party: Principal Investigator, Helena M Verkooijen, Prof.dr., UMC Utrecht
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NL73192.041.20
Record Dates: First submitted 2021-04-22; First posted 2021-04-27 (Actual); Last update posted 2021-08-25 (Actual); Status verified 2021-08

CONDITIONS: Prostate Cancer; Erectile Dysfunction Following Radiation Therapy
MeSH Terms: conditions — Prostatic Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Neurovascular-sparing 5x7.25 Gy MRgRT (Experimental): MRgRT to the prostate in 5 fractions of 7.25 Gy, additionally sparing the neurovascular bundles, internal pudendal arteries, corpora cavernosa, and penile bulb
  Interventions: Radiation: Neurovascular-sparing

INTERVENTIONS:
Radiation: Neurovascular-sparing — Dose reduction of the neurovascular bundles, internal pudendal arteries, corpora cavernosa, and penile bulb during 5x7.25 Gy MRgRT

SUMMARY:
Single-arm phase II trial of 70 men with low- or intermediate-risk prostate cancer receiving magnetic resonance guided adaptive radiotherapy (MRgRT) in 5 fractions of 7.25 Gy, additionally sparing the neurovascular bundles, the internal pudendal arteries, the corpora cavernosa, and the penile bulb for erectile function preservation.

DETAILED DESCRIPTION:
Rationale: Erectile dysfunction is a frequent side effect of external beam radiotherapy (EBRT) for prostate cancer. To date, anatomy-based treatments that are designed to spare relevant neurovascular structures such as the internal pudendal artery and neurovascular bundles have not yet been routinely implemented in clinical practice. The implementation of magnetic resonance imaging (MRI) in treatment planning and introduction of Intensity Modulated Radiotherapy (IMRT) and Volumetric Arc Therapy (VMAT) have improved treatment precision and enabled anatomy-based EBRT and neurovascular-sparing treatments. Spratt et al. have conducted a single-arm phase 2 study to investigate the effect of vascular-sparing IMRT treatments, and found a significantly improved 2-year erectile function (78%, 95% confidence interval [CI] 71-85%) compared to conventional radiotherapy (42%, 95% CI 38-45%; p<0.001) or nerve-sparing prostatectomy (24%, 95% CI 22-27%; p<0.001). In the UMCU, the state-of-the-art MRI linear accelerator (MR-Linac) has recently been introduced. This new system allows radiation delivery under high-precision MRI visualization. The MR-Linac is therefore the most suitable technique for neurovascularsparing external beam radiotherapy treatments. Such neurovascular-sparing treatments may substantially improve post-radiotherapy erectile function outcomes and can thus improve quality of life without substantially compromising oncologic outcome.

Objective: To investigate preservation of erectile function after MR-guided radiotherapy with neurovascular-sparing in patients with localized prostate cancer.

Study design: The EREctile function preservation for prostate Cancer radiation Therapy (ERECT) trial is a prospective, single-center, phase 2 trial. Patients will be treated with the MR-Linac up to 5 fractions of 7.25 Gy with neurovascular-sparing. All fractions will be delivered over the course of 2 and a half weeks.

Study population: Men with low- and intermediate-risk adenocarcinoma of the prostate, clinical stage T1c-T2c, and Gleason ≤7, and iPSA <20 µg/L (NCCN risk categories). Patients with pT1a/b tumor diagnosis after transurethral resection of the prostate (TURP) are included, patients with "bulky" iT3 tumor diagnosis are excluded. Baseline erectile function score according to the International Index of Erectile Function (IIEF-5) questionnaire of at least 17.

Intervention: All patients will receive MR-Linac treatment consisting of 5 fractions of 7.25 Gy with neurovascular sparing, Fractions will be delivered with an overall treatment time of two and a half weeks.

Main study parameters/endpoints:

Primary endpoint: the incidence of erectile dysfunction (ED) three years after treatment.

Secondary endpoints: relapse-free survival, acute and late genitourinary and gastrointestinal toxicity and patient reported quality of life.

Nature and extent of the burden and risks associated with participation, benefit and group relatedness: Participants will receive neurovascular sparing MR guided radiation therapy (MRgRT) consisting of 5 fractions of 7.25 Gy. The number of fractions and duration of treatment is similar to conventional MRgRT consisting of 5 fractions of 7.25 Gy. No increase in toxicity is expected as the dose constraints for the organs at risk in the neurovascular sparing plan will be identical to the conventional plan (i.e. bladder, rectum, femoral head and anal sphincter). For neurovascular sparing treatment, the protocol is extended with dose constraints for newly identified organs at risk (i.e. neurovascular bundles (NVB), internal pudendal arteries (IPA), corpora cavernosa (CC) and penile bulb (PB)). Attention for these organs at risk during treatment planning may reduce erectile dysfunction for the neurovascular sparing treatment. The dose to the dorsolateral part of the prostate might be lower in the NVB sparing plan as the NVB lies in close proximity to this part of the prostate. A slight dose concession on the dorsolateral part of the prostate will only be permitted if the visible tumor on multiparametric MRI is not in vicinity of the NVB as underdosage of the dominant index lesion is undesirable for tumor control. A lower dose to the dorsolateral part of the prostate may have an impact on biochemical control for certain cases, but we do not expect that it will influence overall survival.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥18 years
* Histologically proven adenocarcinoma of the prostate
* Low-risk or intermediate-risk prostate cancer according to NCCN risk categories (low risk: T1c-T2a, Gleason score ≤6, and PSA <10 µg/L; intermediate risk: T2b-T2c or Gleason score 7 or PSA 10-20 µg/L)
* Patients with pT1a/b tumor diagnosis after transurethral resection of the prostate (TURP)
* Domain score of 17-25 on the International Index of Erectile Function-5 (IIEF-5) questionnaire
* Karnofsky score of 70-100
* Written informed consent

Exclusion Criteria:

* Use of (neo-)adjuvant androgen deprivation therapy
* High-risk prostate cancer according to NCCN risk categories (T3a or Gleason score 8-10 or PSA >20 µg/L)
* Patients with "bulky" iT3 tumor diagnosis
* Previous pelvic irradiation or radical prostatectomy
* Clinical evidence of metastatic disease
* Patients who are unable to undergo MRI
* Patients who are incompetent to sign written informed consent

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 70 (Estimated)
Dates: Start 2021-07-14 (Actual); Primary Completion 2025-08-10 (Estimated); Study Completion 2025-08-10 (Estimated)

PRIMARY OUTCOMES:
Erectile dysfuntion | 3 years
  Erectile function score of ≤11 on the International Index of Erectile Function (IIEF) -5 questionnaire (0=worst; 25=best)

SECONDARY OUTCOMES:
Relapse-free survival | 3 years
  Defined as biochemical relapse, or positive PSMA scan or clinical relapse whichever occurs first. Biochemical relapse is defined according to the Phoenix definition, i.e. a PSA greater than the current Nadir plus 2 ng/mL. Clinical relapse consists either of locoregional disease or distant metastases
Patient-reported quality of life | 3 years
  According to the Expanded Prostate Cancer Index Composite short form (EPIC-26) questionnaire
Acute and late gastrointestinal and genitourinary toxicity | 3 years
  According to the Common Terminology Criteria for Adverse Events version 5

CONTACTS AND LOCATIONS:
Overall Officials: Jochem RN van der Voort van Zyp, MD PhD, Principal Investigator — UMC Utrecht
Locations (1):
- University Medical Center Utrecht, Utrecht, Netherlands

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Roy A, Green O, Brenneman R, Bosch W, Gay HA, Michalski JM, Baumann BC. Assessing Inter-Fraction Changes in The Size and Position of The Penile Bulb During Daily MR-Guided Radiation Therapy to The Prostate Bed: Do We Need to Adjust How We Plan Radiation in The Post-Radical Prostatectomy Setting to Reduce Risk of Erectile Dysfunction? Clin Genitourin Cancer. 2022 Jun;20(3):e227-e232. doi: 10.1016/j.clgc.2022.01.006. Epub 2022 Jan 11. PMID 35153154